CLINICAL TRIAL: NCT01310660
Title: Evaluation of Levator Injuries Using Transvaginal Endosonography
Acronym: ELITE
Status: Completed | Type: Observational
Sponsor: Croydon University Hospital (Other)
Responsible Party: Principal Investigator, Ranee Thakar, Consultant Urogynaecologist, Croydon University Hospital
Other Study IDs: 10/H0806/87
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Childbirth Related Levator Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nulliparous

SUMMARY:
Prospective studies to date have identified that the levator ani muscle injuries occur in 14-19% of women after vaginal delivery.

In none of studies a vaginal examination was performed at the time of delivery. It has previously been shown that sonographic injuries of the anal sphincter that were believed to be occult were in fact clinically apparent but not recognised at the time of delivery. It is therefore important to correlate clinical findings to ultrasound images.

3D endovaginal endosonography has not previously been used to identify levator injuries. This should potentially provide a better view of the pelvic floor muscles.

The relationship between levator injury and symptoms of pelvic floor dysfunction has not been previously established using validated questionnaires. In this study, we include validated questionnaires to evaluate urinary incontinence, faecal incontinence and vaginal symptoms. As symptoms may become apparent only in the long term it is prudent that the women are followed up in the long term.

The principle objective is to establish the incidence of levator muscle defects during pregnancy and after childbirth. The levator muscle forms a major part of the pelvic floor and damage to this muscle can potentially cause urinary, bowel and sexual problems and pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women who have not delivered previously
2. Singleton pregnancy
3. Maternal age > 18 years and
4. No previous pregnancies >20 weeks of gestation
5. Ability to read and understand English.

Exclusion Criteria:

1. Pregnant women who have delivered previously
2. Multiple pregnancies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Nulliparous
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The principal objective is to establish the incidence of levator muscle defects during pregnancy and after childbirth. | Antenatal, after delivery and postnatal

CONTACTS AND LOCATIONS:
Locations (1):
- Croydon University Hospital, Croydon, Surrey, United Kingdom